CLINICAL TRIAL: NCT00644631
Title: A Multicenter, Randomized, Parallel Group, Double-Blind, Placebo Controlled, Flexible Dose Escalation Study To Evaluate Sexual And Relationship Satisfaction In The Female Partner Of Men With Erectile Dysfunction Treated With Viagra (Sildenafil Citrate) In The United States
Brief Title: A Multicenter, Randomized, Parallel Group, Double-Blind, Placebo Controlled, Flexible Dose Escalation Study To Evaluate Sexual And Relationship Satisfaction In The Female Partner Of Men With Erectile Dysfunction Treated With Sildenafil Citrate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481177
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg (initial dose) tablet by mouth 30 to 60 minutes prior to sexual activity for 12 weeks; depending upon safety, efficacy and tolerability, the dose could be increased to 100 mg or reduced to 25 mg, if necessary.
  Arms: Arm 1
Drug: placebo — placebo tablet by mouth 30 to 60 minutes prior to sexual activity for 12 weeks
  Arms: Arm 2

SUMMARY:
To compare the effects of sildenafil versus placebo on the female partner's sexual satisfaction as assessed by Question 3 of Female Partner of Erectile Dysfunction (ED) Subject Questionnaire (FePEDS-Q): "Over the past 4 weeks, when you had sexual intercourse, how often was it satisfactory for you?" For ED subjects, determine difference in the Erectile Function domain of International Index of Erectile Function (IIEF) between sildenafil citrate and placebo at end of the treatment phase and determine the overall relationship between improved erectile function and increased ED subject and female partner satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The male patient must have had a documented clinical diagnosis of erectile dysfunction (ED) confirmed by a Sexual Health Inventory-Male (SHI-M) score of less than or equal to 21
* a stable female partner at least 21 years of age for at least 6 months prior to screening
* the couple must have been married or living together at the time of screening.
* The female partner must have answered "no intercourse," "sometimes," "a few times" or "almost never" on Question 3 of the Female Partner of ED Subject Questionnaire (FePEDS-Q)

Exclusion Criteria:

* The male patient must not have had resting sitting and/or standing hypotension (BP < 90/50mmHg) or hypertension (BP > 170/110mmHg), or significant cardiovascular disease in the last 3 months, including cardiac failure, myocardial infarction, unstable angina, stroke, transient ischemic attack (TIA), symptomatic or clinically significant cardiac arrhythmias.
* Female partners must not have had significant dyspareunia or lifelong significant sexual dysfunction based on female partner's medical and sexual history at screening.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-06; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Question 3 of the Female Partner ED Subject Questionnaire (FePEDS-Q) in female partners. | Week 12

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) Erectile Function, Desire, Orgasm, Intercourse Satisfaction, and Overall Satisfaction Domains in ED patients | Week 8 and Week 12
Self-Esteem and Relationship Questionnaire (SEAR) in ED patients | Week 12
ED Subject Event Log in ED patients | Week 12
Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) index of treatment satisfaction in ED patients | Week 12
Dyadic Adjustment Scale (DAS) in ED patients | Week 8 and Week 12
American Urological Association (AUA) Symptom Index in ED patients | Week 12
Global Efficacy Assessment Questions (GEQ) in ED patients | Week 12
Questions 1 and 2 of Female Partner of ED Subject Questionnaire (FePEDS-Q) in female partners | Week 8 and Week 12
Sexual Function Questionnaire (SFQ) Desire, Arousal, Enjoyment and Orgasm Domains in female partners | Week 12
Female Sexual Function Inventory (FSFI) Desire, Satisfaction and Arousal Domains in female partners | Week 12
Partner EDITS in female partners | Week 12
Female Partner Treatment Continuation Question in female partners | Week 12
Dyadic Adjustment Scale (DAS) in female partners | Week 8 and Week 12
Beck Depression Inventory (BDI-II) in female partners | Week 12
Female Partner Event Log in female partners | Week 12
AUA Symptom Index in female partners | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (29):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Peabody, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Newtown, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Lacey, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481177&StudyName=A%20Multicenter%2C%20Randomized%2C%20Parallel%20Group%2C%20Double-Blind%2C%20Placebo%20Controlled%2C%20Flexible%20Dose%20Escalation%20Study%20To%20Evaluate%20Sexual%20And%20R